CLINICAL TRIAL: NCT03681912
Title: Tailored Motivational Interviewing Implementation-Effectiveness Trial in Multidisciplinary Adolescent HIV Care Settings
Acronym: TMI
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Collaborators: St. Jude Children's Research Hospital (Other); Children's Hospital of Philadelphia (Other); State University of New York (Other); University of Miami (Other); Johns Hopkins University (Other); University of California, San Diego (Other); University of Alabama at Birmingham (Other); University of South Florida (Other); Children's Hospital Los Angeles (Other); Children's National Research Institute (Other); City University of New York, School of Public Health (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Sylvie Naar, Principal Investigator, Florida State University
Other Study IDs: ATN 146
Record Dates: First submitted 2018-09-07; First posted 2018-09-24 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections; Adolescent Development; Care Eliciting Behavior; Patient Non-Compliance; Patient Refusal of Treatment
Keywords: Implementation Science; Motivational Interviewing; Youth Living with HIV
MeSH Terms: conditions — HIV Infections; Patient Compliance; Treatment Refusal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (15):
- Implementation Block 1: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 3 months.
  Interventions: Behavioral: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS)
- Implementation Block 2: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 6 months.
  Interventions: Behavioral: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS)
- Implementation Block 3: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 9 months.
  Interventions: Behavioral: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS)
- Implementation Block 4: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 12 months.
  Interventions: Behavioral: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS)
- Implementation Block 5: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 15 months.
  Interventions: Behavioral: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS)
- Sustainment Block 1 Facilitated CoP: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
  Interventions: Behavioral: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
- Sustainment Block 2 Facilitated CoP: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
  Interventions: Behavioral: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
- Sustainment Block 3 Facilitated CoP: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
  Interventions: Behavioral: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
- Sustainment Block 4 Facilitated CoP: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
  Interventions: Behavioral: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
- Sustainment Block 5 Facilitated CoP: Randomized Guided Development of CoPs with an internal facilitator after one year of implementation.
  Interventions: Behavioral: Randomized Guided Development of COPs with an internal facilitator after one year of implementation.
- Sustainment Block 1 CoP Alone: After one year of implementation, site is randomized to receive CoP development without internal facilitation.
  Interventions: Behavioral: CoP development without internal facilitation.
- Sustainment Block 2 CoP Alone: After one year of implementation, site is randomized to receive CoP development without internal facilitation.
  Interventions: Behavioral: CoP development without internal facilitation.
- Sustainment Block 3 CoP Alone: After one year of implementation, site is randomized to receive CoP development without internal facilitation.
  Interventions: Behavioral: CoP development without internal facilitation.
- Sustainment Block 4 CoP Alone: After one year of implementation, site is randomized to receive CoP development without internal facilitation.
  Interventions: Behavioral: CoP development without internal facilitation.
- Sustainment Block 5 CoP Along: After one year of implementation, site is randomized to receive CoP development without internal facilitation.
  Interventions: Behavioral: CoP development without internal facilitation.

INTERVENTIONS:
Behavioral: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) — Coaching feedback will be triggered by a provider falling below the competency threshold on the standardized patient interaction. Everyone will receive coaching for two assessments in the month following training. After that, if mean scores fall below competency, then the provider will receive a 45-minute coaching session by the external Motivational Interviewing Network of Trainers (MINT) facilitator.
  Feedback on two highest and two lowest ratings, review of the audio recording and interactive coaching activities (e.g., fidelity assessments) targeting the lowest ratings. While many aspects of this implementation strategy are adaptable, organizational leadership will review data on completion of coaching feedback sessions and will determine corrective action for suboptimal adherence.
  Groups: Implementation Block 1; Implementation Block 2; Implementation Block 3; Implementation Block 4; Implementation Block 5
Behavioral: Randomized Guided Development of COPs with an internal facilitator after one year of implementation. — Development of the CoP will be guided by scheduling and assisting in setting the agenda for the first three meetings to encourage MI practice, peer coaching and potentially fidelity monitoring, and prevent drift. In addition to CoP, half the sites will be randomized to receive an internal facilitator who will be trained to continue quarterly fidelity monitoring and coaching feedback when scores fall below competency.
  Groups: Sustainment Block 1 Facilitated CoP; Sustainment Block 2 Facilitated CoP; Sustainment Block 3 Facilitated CoP; Sustainment Block 4 Facilitated CoP; Sustainment Block 5 Facilitated CoP
Behavioral: CoP development without internal facilitation. — Development of the CoP will be guided by scheduling and assisting in setting the agenda for the first three meetings to encourage MI practice, peer coaching and potentially fidelity
  Groups: Sustainment Block 1 CoP Alone; Sustainment Block 2 CoP Alone; Sustainment Block 3 CoP Alone; Sustainment Block 4 CoP Alone; Sustainment Block 5 CoP Along

SUMMARY:
The goal of this study is to test a multi-faceted Tailored Motivational Interviewing Implementation intervention (TMI), based on the Dynamic Adaptation Process (DAP) to scale up an Evidence-based Practice (EBP) in multidisciplinary adolescent HIV care settings while balancing flexibility and fidelity.

A mixed-methods design will be used, in which the dominant method is quantitative (a dynamic wait-listed design; DWLD) to determine the impact of TMI on the integration of MI with fidelity in 10 adolescent HIV clinics with an average of 15 providers and 100 patients each.

DETAILED DESCRIPTION:
The NIH Office of AIDS Research called for implementation science (IS) to address the behavioral research-practice gap.Motivational Interviewing (MI) is the only behavioral intervention to date shown to be effective to improve self-management for youth living with HIV (YLH). MI was also the only intervention to demonstrate success across the youth HIV care cascade. MI interventions can target multiple behaviors and be delivered by multiple provider-types as is common in adolescent HIV care settings. Finally, MI is already embedded in the clinical guidelines for HIV care and HIV risk reduction. Implementation Science is the scientific study of methods to promote the uptake of research findings and evidence-based practice (EBPs) to improve the quality of behavior change approaches in health care settings. A primary challenge of scaling up EBP's is the balance of flexibility (adaptation to context) and fidelity (provider adherence and competence). The Dynamic Adaptation Process (DAP) guides tailoring of MI implementation at the exploration, preparation, implementation, and sustainment phases (EPIS) of scale up. The goal of this proposal is to test a multi-faceted Tailored Motivational Interviewing, Implementation intervention (TMI), based on the DAP to scale up an EBP in multidisciplinary adolescent HIV care settings while balancing flexibility and fidelity.

The pilot work for TMI included tailoring of initial workshop training based on innovative methods in communication science, developing efficient fidelity measurement, and pilot testing the revised intervention. The initial TMI workshop was adapted based on findings from sequential analysis of provider interactions with youth living with HIV (YLH) by emphasizing provider communication strategies most associated with patient motivational statements ("change talk"), de-emphasizing MI strategies that were unrelated to change talk, and suppressing those that were associated with a motivational statements ("counter-change talk"). Additional tailoring based on the DAP requires that qualitative and quantitative data are collected during the exploration phase. In the preparation phase, these data are reviewed by an implementation team comprised of local stakeholders and experts in MI implementation who recommend necessary adaptations for the service context while balancing the need for fidelity (adherence to minimum implementation requirements and achieving provider competency thresholds). In the implementation phase, ongoing fidelity monitoring determines the need for ongoing coaching, thus amount of coaching is tailored to the individual provider. Finally, the sustainment phase addresses the maintenance of innovation beyond 1 year utilizing strategies such as developing communities of practice (CoPs) and promoting internal facilitation of TMI.

In a hybrid implementation-effectiveness (Type 3) trial, the effect of TMI will be tested on fidelity EBP, and secondarily on HIV cascade-related outcomes, using a dynamic wait-listed design (DWLD) 18 with 165 providers nested within 10 Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN4) sites. With this design, the 10 clinics will be randomly assigned in 5 clusters to receive TMI. For each randomization, 2 clinics receive TMI and the others remain in the wait-list condition. This will continue until the 5th cluster has been randomized to TMI. After one year of TMI's external facilitation based on the DAP, a second randomization will compare internal facilitator monitoring and coaching plus the encouragement of CoPs to CoPs alone. Fidelity will be assessed on a quarterly basis through the 24 months of intervention and an additional 6 months of follow-up. The proposal uses the EPIS model, to guide the investigation of the interacting elements that influence successful implementation. The qualitative method will be nested within the quantitative study to provide a deeper understanding of the implementation context and understand why or why not MI is integrated with fidelity across the 150 providers. Providers and key stakeholders will complete qualitative interviews and brief assessments based on EPIS at baseline, after one year of TMI (first randomization), and after 1 year of follow-up (second randomization).

ELIGIBILITY:
Inclusion Criteria:

* All youth HIV providers (prevention and care) at our target clinics will be eligible to participate.

Exclusion Criteria:

* Non-providers of youth HIV prevention and care

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Providers of prevention and care for youth with HIV
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Todd, MS, JD, Study Chair — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Coyle K, Carcone AI, Butame S, Pooler-Burgess M, Chang J, Naar S. Adapting the self-assessment of contextual fit scale for implementation of evidence-based practices in adolescent HIV settings. Implement Sci Commun. 2022 Oct 22;3(1):115. doi: 10.1186/s43058-022-00349-4. PMID 36273221
- [Derived] Naar S, MacDonell K, Chapman JE, Todd L, Gurung S, Cain D, Dilones RE, Parsons JT. Testing a Motivational Interviewing Implementation Intervention in Adolescent HIV Clinics: Protocol for a Type 3, Hybrid Implementation-Effectiveness Trial. JMIR Res Protoc. 2019 Jun 7;8(6):e11200. doi: 10.2196/11200. PMID 31237839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: TMI study staff will work with the SC at each site to introduce the project and recruit participants by scheduling and conducting introductory meetings. After the introductory meetings, the SC or PI from each site will send contact information (email, phone number) to the TMI study staff. The TMI study staff will contact participants via email and/or phone call to provide the information sheet and schedule of assessments.
Units Other Than Participants: Site
Groups:
- Block 1 Site 7: Site 7 was randomized into Block 1 at baseline. In our stepped wedged design, this site entered the implementation phase first, along with site 10, and randomized at the sustainment phase.
- Block 1 Site 10: Site 10 was randomized into Block 1 at baseline. In our stepped wedged design, this site entered the implementation phase first, along with site 7, and randomized at the sustainment phase.
- Block 2 Site 3: Site 3 was randomized into Block 2 at baseline. In our stepped wedged design, this site entered the implementation phase second, along with site 8, and randomized at the sustainment phase.
- Block 2 Site 8: Site 8 was randomized into Block 2 at baseline. In our stepped wedged design, this site entered the implementation phase second, along with site 3, and randomized at the sustainment phase.
- Block 3 Site 1: Site 1 was randomized into Block 3 at baseline. In our stepped wedged design, this site entered into implementation phase third, along with Site 11, and randomized at the sustainment phase.
- Block 3 Site 11: Site 11 was randomized into Block 3 at baseline. In our stepped wedged design, this site entered the implementation phase third, along with site 1, and randomized at the sustainment phase.
- Block 4 Site 2: Site 2 was randomized into Block 4 at baseline. In our stepped wedged design, this site entered the implementation phase fourth, along with site 12, and randomized at the sustainment phase.
- Block 4 Site 12: Site 12 was randomized to Block 4 at baseline. In our stepped wedged design, this site entered the implementation phase fourth, along with Site 2, and randomized at the sustainment phase.
- Block 5 Site 6: Site 6 was randomized into Block 5 at baseline. In our stepped wedged design, this site entered the implementation phase fifth, along with site 13, and randomized at the sustainment phase.
- Block 5 Site 13: Site 13 was randomized into Block 5 at baseline. In our stepped wedged design, this site entered the implementation phase fifth, along with site 6, and randomized at the sustainment phase.
Period: Overall Study
Arm/Group | Block 1 Site 7 | Block 1 Site 10 | Block 2 Site 3 | Block 2 Site 8 | Block 3 Site 1 | Block 3 Site 11 | Block 4 Site 2 | Block 4 Site 12 | Block 5 Site 6 | Block 5 Site 13
Started | 18; 1 Site | 11; 1 Site | 18; 1 Site | 16; 1 Site | 17; 1 Site | 15; 1 Site | 19; 1 Site | 24; 1 Site | 28; 1 Site | 22; 1 Site
Completed | 14; 1 Site | 8; 1 Site | 7; 1 Site | 8; 1 Site | 9; 1 Site | 10; 1 Site | 11; 1 Site | 14; 1 Site | 12; 1 Site | 13; 1 Site
Not Completed | 4; 0 Site | 3; 0 Site | 11; 0 Site | 8; 0 Site | 8; 0 Site | 5; 0 Site | 8; 0 Site | 10; 0 Site | 16; 0 Site | 9; 0 Site

BASELINE CHARACTERISTICS:
Groups:
- Block 1 Site 7; Block 1 Site 10; Block 2 Site 3; Block 2 Site 8; Block 3 Site 1; Block 3 Site 11; Block 4 Site 2; Block 4 Site 12; Block 5 Site 6; Block 5 Site 13: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 3 months.
- Total: Total of all reporting groups
Arm/Group | Block 1 Site 7 | Block 1 Site 10 | Block 2 Site 3 | Block 2 Site 8 | Block 3 Site 1 | Block 3 Site 11 | Block 4 Site 2 | Block 4 Site 12 | Block 5 Site 6 | Block 5 Site 13 | Total
Number analyzed (Participants) | 18 | 11 | 18 | 16 | 17 | 15 | 19 | 24 | 28 | 22 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 11 | 18 | 16 | 17 | 15 | 19 | 24 | 28 | 22 | 188
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 17 | 8 | 14 | 11 | 9 | 9 | 12 | 5 | 6 | 7 | 98
  Female | 0 | 2 | 2 | 2 | 1 | 2 | 1 | 3 | 4 | 0 | 17
  Unknown | 1 | 1 | 2 | 3 | 7 | 4 | 6 | 16 | 18 | 15 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Black / African American | 9 | 1 | 3 | 6 | 6 | 4 | 7 | 3 | 8 | 4 | 51
  Middle Eastern / North African | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 7 | 7 | 12 | 5 | 4 | 9 | 7 | 3 | 2 | 2 | 58
  Other | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 6
  Unknown | 1 | 1 | 2 | 3 | 7 | 2 | 5 | 15 | 18 | 15 | 69
  Hispanic | 0 | 5 | 6 | 2 | 0 | 1 | 0 | 4 | 0 | 1 | 19
  Not Hispanic | 17 | 5 | 10 | 11 | 10 | 12 | 14 | 5 | 10 | 6 | 100
  Uknown Hispanic | 1 | 1 | 2 | 3 | 7 | 2 | 5 | 15 | 18 | 15 | 69
Motivational Interviewing (MI) Coach Rating Scale (CRS) (Raw Average) [Mean (Standard Deviation); unit: Units on a scale] — Motivational Interviewing (MI) Coach Rating Scale (CRS) is a 12-item measure, rated on a 4-point categorical rating scale (1=Poor, 2=Fair, 3=Good, 4=Excellent). A coder selected a 15 minute portion of the session and coded the provider's MI skills (e.g., empathy, collaboration, supporting autonomy, open ended questions, etc.). The 12 items were averaged with a min of 1 and max of 4. The final competence categories were: Beginner (<2.0), Novice (>=2.0 and <2.6), Intermediate (>=2.6 and <3.3), and Advanced (>=3.3), analyzed according to a Gaussian distribution.
  Units on a scale | 2.21 (0.44) | 1.99 (0.24) | 1.77 (0.26) | 1.80 (0.36) | 1.92 (0.34) | 2.36 (0.41) | 1.98 (0.42) | 1.77 (0.32) | 1.92 (0.35) | 2.03 (0.36) | 1.96 (0.39)
Motivational Interviewing (MI) Coach Rating Scale (CRS) Criterion Score [Mean (Standard Deviation); unit: Units on a scale] — Motivational Interviewing (MI) Coach Rating Scale (CRS) is a 12-item measure, rated on a 4-point categorical rating scale (1=Poor, 2=Fair, 3=Good, 4=Excellent). A coder selected a 15 minute portion of the session and coded the provider's MI skills (e.g., empathy, collaboration, supporting autonomy, open ended questions, etc.). The 12 items were averaged with a min of 1 and max of 4. The final competence categories were: Beginner (<2.0), Novice (>=2.0 and <2.6), Intermediate (>=2.6 and <3.3), and Advanced (>=3.3), analyzed according to an ordinal distribution (logit link).
  Units on a scale | 1.89 (0.68) | 1.50 (0.50) | 1.28 (0.34) | 1.33 (0.47) | 1.39 (0.52) | 2.06 (0.66) | 1.63 (0.69) | 1.33 (0.48) | 1.46 (0.52) | 1.58 (0.52) | 1.53 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Raw Average: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS)
Description: Providers will complete a 15-minute standard patient role-play at each point during baseline, implementation and sustainment.
  The Research Assistant (RA) will code these interactions on the 12-item MI CRS and reliability will continue to be monitored with one coding per month co-coded by Dr. Naar. These reports will be cumulatively reported and collected quarterly. Each item on the CRS has a score of 1 (lowest) to 4 (highest). The 12 scores are added and averaged for a score that reflects competency: <2.0=Beginner. >=2.0 to <2.6. >=2.6 to <3.3=Intermediate. >=3.3=Advanced. The outcomes provided below represent the average of the provider scores and reported by site and implementation phase.
  For sites randomized to internal facilitation in the sustainment period, the RA will code the same interactions so that the facilitator ratings will not be used for research purposes.
Time Frame: Every three months over fifteen months
Population: Participants may choose to leave the study at any point. Participants may be removed from the study based on changes in their clinical role and if they have less than 4 hours of client contact per week on average. Participant data will be included, unless a participant requests that their data is removed. In such cases, the participant's data will be deleted.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Block 1 Site 7 - CoP Alone; Block 2 Site 8 - CoP Alone; Block 3 Site 11 - CoP Alone; Block 4 Site 12 - CoP Alone; Block 5 Site 6 - CoP Alone: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS): Coaching feedback will be triggered by a provider falling below the competency threshold on the standardized patient interaction. Everyone will receive coaching for two assessments in the month following training. After that, if mean scores fall below competency, then the provider will receive a 45-minute coaching session by the external Motivational Interviewing Network of Trainers (MINT) facilitator.
  Feedback on two highest and two lowest ratings, review of the audio recording and interactive coaching activities (e.g., fidelity assessments) targeting the lowest ratings. While many aspects of this implementation strategy are adaptable, organizational leadership will review data on completion of coaching feedback sessions and will determine corrective action for suboptimal adherence.
  CoP development without internal facilitation.: Development of the CoP will be guided by scheduling and assisting in setting the agenda for the first three meetings to encourage MI practice, peer coaching and potentially fidelity
- Block 1 Site 10 - CoP Facilitated; Block 2 Site 3 - CoP Facilitated; Block 3 Site 1 - CoP Facilitated; Block 4 Site 2 - CoP Facilitated; Block 5 Site 13 - CoP Facilitated: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS): Coaching feedback will be triggered by a provider falling below the competency threshold on the standardized patient interaction. Everyone will receive coaching for two assessments in the month following training. After that, if mean scores fall below competency, then the provider will receive a 45-minute coaching session by the external Motivational Interviewing Network of Trainers (MINT) facilitator.
  Feedback on two highest and two lowest ratings, review of the audio recording and interactive coaching activities (e.g., fidelity assessments) targeting the lowest ratings. While many aspects of this implementation strategy are adaptable, organizational leadership will review data on completion of coaching feedback sessions and will determine corrective action for suboptimal adherence.
  Randomized Guided Development of COPs with an internal facilitator after one year of implementation.: Development of the CoP will be guided by scheduling and assisting in setting the agenda for the first three meetings to encourage MI practice, peer coaching and potentially fidelity monitoring, and prevent drift. In addition to CoP, half the sites will be randomized to receive an internal facilitator who will be trained to continue quarterly fidelity monitoring and coaching feedback when scores fall below competency.
Arm/Group | Block 1 Site 7 - CoP Alone | Block 1 Site 10 - CoP Facilitated | Block 2 Site 3 - CoP Facilitated | Block 2 Site 8 - CoP Alone | Block 3 Site 1 - CoP Facilitated | Block 3 Site 11 - CoP Alone | Block 4 Site 2 - CoP Facilitated | Block 4 Site 12 - CoP Alone | Block 5 Site 6 - CoP Alone | Block 5 Site 13 - CoP Facilitated
Number analyzed (Participants) | 16 | 10 | 13 | 13 | 11 | 12 | 13 | 19 | 17 | 17
Units on a scale
  Implementation Phase | 2.72 (0.45) | 2.50 (0.46) | 1.99 (0.34) | 2.32 (0.51) | 2.47 (0.53) | 2.91 (0.37) | 2.62 (0.50) | 2.39 (0.43) | 2.63 (0.49) | 2.66 (0.48)
  Sustainment Phase: number analyzed (Participants) | 14 | 8 | 7 | 8 | 9 | 10 | 11 | 14 | 12 | 13
  Sustainment Phase | 2.78 (0.43) | 2.59 (0.26) | 2.19 (0.37) | 2.19 (0.26) | 2.38 (0.56) | 2.82 (0.43) | 2.73 (0.51) | 2.41 (0.48) | 2.76 (0.61) | 2.65 (0.45)

2. Secondary Outcome: Change in Individual Patients' Records Report Related to HIV Viral Load
Description: Record/chart abstraction conducted for patients in care at the site for
  * The 12 months prior to the start of implementation
  * The 12 months during implementation; and
  * The 6 months after the end of the implementation intervention.
  These data include viral load
Time Frame: 12 months prior to start; The end of the 12 month intervention, and 6 months after end of implementation interview
Population: Record/Chart Abstraction was conducted based on number of patients at clinic for a given year. Clinic patient population numbers fluctuate.
Measure: Mean (Standard Deviation); unit: Log of copies/mL
Groups:
- Block 1 Site 7; Block 2 Site 8; Block 3 Site 11; Block 4 Site 12; Block 5 Site 6: Communities of Practice (CoP) development without internal facilitation.
- Block 1 Site 10; Block 2 Site 3; Block 3 Site 1; Block 4 Site 2; Block 5 Site 13: Randomized Guided Development of Communities of Practice (CoP) with an internal facilitator after one year of implementation.
Arm/Group | Block 1 Site 7 | Block 1 Site 10 | Block 2 Site 3 | Block 2 Site 8 | Block 3 Site 1 | Block 3 Site 11 | Block 4 Site 2 | Block 4 Site 12 | Block 5 Site 6 | Block 5 Site 13
Number analyzed (Participants) | 246 | 91 | 146 | 78 | 186 | 144 | 124 | 206 | 130 | 111
Log of copies/mL
  Baseline Phase - 12 months prior to the start of implementation | 1.88 (0.80) | 2.43 (1.04) | 2.29 (1.05) | 2.28 (1.12) | 2.30 (1.17) | 2.20 (0.99) | 2.36 (1.25) | 2.35 (1.20) | 1.92 (1.70) | 1.11 (2.89)
  Implementation Phase - 12 months during implementation: number analyzed (Participants) | 218 | 62 | 105 | 63 | 172 | 107 | 78 | 85 | 58 | 66
  Implementation Phase - 12 months during implementation | 1.85 (0.86) | 1.81 (0.61) | 2.12 (1.25) | 1.89 (0.97) | 2.00 (1.07) | 2.07 (1.09) | 2.12 (1.27) | 2.10 (1.21) | 1.78 (1.49) | 2.38 (1.25)
  Sustainment Phase - 6 months after the end of the implementation: number analyzed (Participants) | 230 | 66 | 92 | 68 | 186 | 84 | 107 | 56 | 43 | 51
  Sustainment Phase - 6 months after the end of the implementation | 1.88 (0.83) | 1.80 (0.59) | 2.31 (1.23) | 2.00 (1.10) | 1.98 (1.08) | 1.90 (0.77) | 2.22 (1.19) | 1.76 (0.87) | 1.79 (0.77) | 2.17 (1.15)

ADVERSE EVENTS:
Time Frame: Not applicable as we did not monitor for adverse events.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed because the study was deemed no more than minimal risk.
Groups:
- Implementation Block 1: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 3 months.
  Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS): Coaching feedback will be triggered by a provider falling below the competency threshold on the standardized patient interaction. Everyone will receive coaching for two assessments in the month following training. After that, if mean scores fall below competency, then the provider will receive a 45-minute coaching session by the external Motivational Interviewing Network of Trainers (MINT) facilitator.
  Feedback on two highest and two lowest ratings, review of the audio recording and interactive coaching activities (e.g., fidelity assessments) targeting the lowest ratings. While many aspects of this implementation strategy are adaptable, organizational leadership will review data on completion of coaching feedback sessions and will determine corrective action for suboptimal adherence.
- Implementation Block 2: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 6 months.
  Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS): Coaching feedback will be triggered by a provider falling below the competency threshold on the standardized patient interaction. Everyone will receive coaching for two assessments in the month following training. After that, if mean scores fall below competency, then the provider will receive a 45-minute coaching session by the external Motivational Interviewing Network of Trainers (MINT) facilitator.
  Feedback on two highest and two lowest ratings, review of the audio recording and interactive coaching activities (e.g., fidelity assessments) targeting the lowest ratings. While many aspects of this implementation strategy are adaptable, organizational leadership will review data on completion of coaching feedback sessions and will determine corrective action for suboptimal adherence.
- Implementation Block 3: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 9 months.
  Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS): Coaching feedback will be triggered by a provider falling below the competency threshold on the standardized patient interaction. Everyone will receive coaching for two assessments in the month following training. After that, if mean scores fall below competency, then the provider will receive a 45-minute coaching session by the external Motivational Interviewing Network of Trainers (MINT) facilitator.
  Feedback on two highest and two lowest ratings, review of the audio recording and interactive coaching activities (e.g., fidelity assessments) targeting the lowest ratings. While many aspects of this implementation strategy are adaptable, organizational leadership will review data on completion of coaching feedback sessions and will determine corrective action for suboptimal adherence.
- Implementation Block 4: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 12 months.
  Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS): Coaching feedback will be triggered by a provider falling below the competency threshold on the standardized patient interaction. Everyone will receive coaching for two assessments in the month following training. After that, if mean scores fall below competency, then the provider will receive a 45-minute coaching session by the external Motivational Interviewing Network of Trainers (MINT) facilitator.
  Feedback on two highest and two lowest ratings, review of the audio recording and interactive coaching activities (e.g., fidelity assessments) targeting the lowest ratings. While many aspects of this implementation strategy are adaptable, organizational leadership will review data on completion of coaching feedback sessions and will determine corrective action for suboptimal adherence.
- Implementation Block 5: Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS) performed monthly but reported quarterly, starting at 15 months.
  Competency: 12-Item Motivational Interviewing (MI) Coach Rating Scale (CRS): Coaching feedback will be triggered by a provider falling below the competency threshold on the standardized patient interaction. Everyone will receive coaching for two assessments in the month following training. After that, if mean scores fall below competency, then the provider will receive a 45-minute coaching session by the external Motivational Interviewing Network of Trainers (MINT) facilitator.
  Feedback on two highest and two lowest ratings, review of the audio recording and interactive coaching activities (e.g., fidelity assessments) targeting the lowest ratings. While many aspects of this implementation strategy are adaptable, organizational leadership will review data on completion of coaching feedback sessions and will determine corrective action for suboptimal adherence.
Arm/Group | Implementation Block 1 | Implementation Block 2 | Implementation Block 3 | Implementation Block 4 | Implementation Block 5 | Sustainment Block 1 Facilitated CoP | Sustainment Block 2 Facilitated CoP | Sustainment Block 3 Facilitated CoP | Sustainment Block 4 Facilitated CoP | Sustainment Block 5 Facilitated CoP | Sustainment Block 1 CoP Alone | Sustainment Block 2 CoP Alone | Sustainment Block 3 CoP Alone | Sustainment Block 4 CoP Alone | Sustainment Block 5 CoP Along
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03681912/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03681912/SAP_001.pdf